CLINICAL TRIAL: NCT04217200
Title: Pregnancy Dating Test - The Fall of hPL in Urine Over Time
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Anatole S Menon-Johansson, Deputy Clinical Lead, Sexual & Reproductive Health Department, Guy's and St Thomas' NHS Foundation Trust
Other Study IDs: IRAS 198143
Record Dates: First submitted 2018-08-16; First posted 2020-01-03 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Abortion, Complete; Miscarriage Threatening
MeSH Terms: conditions — Abortion, Threatened

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Earlier studies describe the half-life of hPL in serum as being ninety minutes and that the hormone is excreted unchanged in urine; consequently, there is real potential to use the fall in hormone levels in urine to monitor bleeding in pregnancy, the outcome of natural and artificial abortions or placental health.

This study will focus on the fall of hPL following delivery by Caesarean section when women have a urinary catheter in place and sampling urine is simple to achieve.

DETAILED DESCRIPTION:
The hormone hPL has a 90 minute half life in serum and the consequently since it is excreted unchanged in the urine it could be a useful marker to evaluate bleeding in pregnancy, determine if a pregnancy has ended by natural and artificial abortion or if there has been a change in placental function during a normal pregnancy.

The project will recruit twelve pregnant women having an elective Caesarean section to determine the fall in hPL over time. Urine samples will be taken just prior to and then every 30 minutes for the first six hours after delivery by Caesarean section.

Pregnant women presenting for an elective Caesarean section at Guy's & St Thomas' NHS Foundation Trust (GSTFT) will be approached to join this study and the following will be done:

1. Invited to participate in study and given Patient Information Leaflet
2. Informed consent obtained
3. Eligibility for inclusion determined
4. A urine sample (20ml) will be collected prior to the Caesarean from the urinary catheter
5. Then urine samples (20mls) will be collected every 30 minutes for the first six hours following Caesarean section delivery
6. The result of the dating ultrasound scan will be added to the trial documentation record
7. The weight of the baby will be added to the trial documentation record

Consent The patient information leaflet clearly states the purpose of the research and the low risk of participation. The co-signing researcher on the consent form will ensure that the signee understands the alternative, is able to retain the relevant information, has capacity and is exercising free choice.

Risks, burdens and benefits This trial involves the collection of serial urine samples. The clinical history and result of the dating ultrasound scan will be recorded to estimate the gestation at delivery. The analysis of these samples will have no bearing on their clinical care.

Confidentiality All women recruited to the trial will be given a unique trial number. The trial data sheet will have the following information. The trial site, unique trial number, date of birth, date, estimated gestation from the result from the dating ultrasound scan. The samples collected will have the following information recorded: the unique trial number, date of birth, date and trial site code.

Conflict of interest None has been identified.

Use of tissue samples in future research The samples will not be stored.

ELIGIBILITY:
Inclusion Criteria:

1. The women is 18 years of age or older
2. She understands the patient information leaflet, trial requirements and has signed the consent form
3. The Caesarean delivery will be at GSTFT
4. Prepared for urine to be collected for up to when the urinary catheter is removed or six hours, whichever is sooner
5. Agrees for the demographic and medical history data to be collected.

Exclusion Criteria:

1. Under 18 years of age
2. Unable to understand the patient information leaflet or consent to join the trial
3. The Caesarean delivery will not be at GSTFT
4. The women is not for urine to be collected
5. The women does not agree for demographic or history data to be collected.
6. The women has a haemorrhage greater than one litre during the Caesarean delivery

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with a singleton pregnancy presenting for a Caesarean section delivery
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
The rate of change in human placental lactogen concentration in urine post delivery by Caesarian section | Baseline and then 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330 & 360 minutes after delivery of the baby by Caesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Anatole S Menon-Johansson, PhD,MPH,FRCP, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All samples will be labelled with a trial identifier when they are sent to the laboratory for analysis. Only the PI will know the link between the trial identifier and the patient clinic number. The patient clinic number can only be linked to an identifiable patient by staff who have access to the hospital electronic patient record.

REFERENCES:
- [Result] Whittaker PG, Lind T, Lawson JY. A prospective study to compare serum human placental lactogen and menstrual dates for determining gestational age. Am J Obstet Gynecol. 1987 Jan;156(1):178-82. doi: 10.1016/0002-9378(87)90233-x. PMID 3541617